CLINICAL TRIAL: NCT02876510
Title: Phase I Adoptive Cellular Therapy Trial With Endogenous CD8+ T Cells (ACTolog® IMA101) Alone or in Combination With Atezolizumab in Patients With Relapsed and/or Refractory Solid Cancers
Brief Title: ACTolog in Patients With Solid Cancers
Acronym: ACTolog
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Immatics US, Inc. (Industry)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMA101-101
Record Dates: First submitted 2016-08-08; First posted 2016-08-23 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Cancer; Solid Tumor
Keywords: Ovarian Cancer; Esophageal Cancer; Head and neck squamous cell carcinoma; non-small cell lung cancer; Gastric Cancer; T-cell Therapy; immunotherapy; adoptive cellular therapy; T-cell receptor; cell therapy; cytotherapy; IMA101; atezolizumab; Tecentriq
MeSH Terms: conditions — Neoplasms; Ovarian Neoplasms; Esophageal Neoplasms; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Non-Small-Cell Lung; Stomach Neoplasms | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; aldesleukin; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- IMA101 product only (Cohort 1) (Experimental): * Pre-conditioning by non-myeloablative chemotherapy with Fludarabine and Cyclophosphamide
  * Infusion of the IMA101 T-cell product(s)
  * Post-infusion administration of low-dose recombinant human interleukin-2
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: IMA101 product; Biological: Recombinant human interleukin-2; Diagnostic Test: IMADetect
- IMA101 product + atezolizumab (Cohort 2) (Experimental): * Pre-conditioning by non-myeloablative chemotherapy with Fludarabine and Cyclophosphamide
  * Infusion of the IMA101 T-cell product(s)
  * Post-infusion administration of low-dose recombinant human interleukin-2
  * Treatment with atezolizumab every 3 weeks after IMA101 product infusion, for 1 year
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: IMA101 product; Biological: Recombinant human interleukin-2; Diagnostic Test: IMADetect; Drug: Atezolizumab

INTERVENTIONS:
Drug: Fludarabine — Fludarabine infusion
  Other Names: Fludarabine monophosphate
Drug: Cyclophosphamide — Cyclophosphamide infusion
  Other Names: Cytoxan
Biological: IMA101 product — i.v. infusion of IMA101 product(s).
Biological: Recombinant human interleukin-2 — Low dose IL-2 Infusion for two weeks
  Other Names: Aldesleukin; Proleukin
Diagnostic Test: IMADetect — IMADetect is a laboratory test that is part of screening used to determine the mRNA expression of ACTolog target source genes in tumor biopsies from solid tumors. IMADetect is intended for investigational use only.
Drug: Atezolizumab — Atezolizumab infusion will be given no earlier than 3 weeks post IMA101 infusion and after hematologic recovery is achieved, thereafter every 3 weeks until 1 year after IMA101 infusion.
  Other Names: Tecentriq
  Arms: IMA101 product + atezolizumab (Cohort 2)

SUMMARY:
The study purpose is to learn about the safety and tolerability of IMA101 alone (Cohort 1) or in combination with atezolizumab (Cohort 2) in patients with advanced solid cancers that express pre-defined Immatics tumor targets.

DETAILED DESCRIPTION:
SCREENING: Patient eligibility will be determined by HLA (human leukocyte antigen) and the main biomarkers screening. If the patient is eligible, white blood cells will be collected with a leukapheresis for the manufacture of the IMA101 product.

MANUFACTURE: IMA101 product will be made from the patient's white blood cells.

TREATMENT: IMA101 product will be administered to the patient intravenously after lymphodepleting pre-conditioning with chemotherapy (fludarabine and cyclophosphamide).

Low-dose IL-2 will be self-administered twice daily for a total of 28 doses after infusion of IMA101 product. In Cohort 2, atezolizumab will be administered every 3 weeks, starting no earlier than 3 weeks after the IMA101 product infusion and after hematologic recovery.

Patients will be monitored closely throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have pathologically confirmed advanced/metastatic cancer prior to enrollment.
2. HLA phenotype positive.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
4. Life expectancy > 6 months prior to enrollment.
5. Patient is a candidate for a maximum of one further line of established therapy (prior to treatment with ACTolog).
6. The patient has adequate organ and marrow function per protocol
7. At least one lesion (metastasis or primary tumor) being considered accessible by non-high-risk collection procedures for biopsy.
8. The patient has adequate hepatic function per protocol
9. The patient has serum creatinine clearance ≥50 mL/min by the Cockcroft-Gault formula.
10. The patient has adequate pulmonary function per protocol
11. Acceptable coagulation status
12. Women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.
13. Male subjects must agree to use effective contraception or abstinence while on study and for 90 days after infusion of the ACTolog T-cell product.
14. Ability of subject to understand and the willingness to sign written informed consent for study participation.
15. Confirmed availability of production capacities for the patient's ACTolog products.
16. ACTolog target expression as evaluated by the in vitro diagnostic device IMA_Detect: Patient's tumor must express at least one ACTolog target as assessed by quantitative PCR (qPCR) (to be assessed from a tumor biopsy to be performed if all other eligibility criteria are met).

Exclusion Criteria

1. Any condition contraindicating leukapheresis.
2. Patients with brain metastases. Patients with a history of brain metastases may be eligible, if an imaging scan with contrast enhancement not older than 4 weeks is able to exclude the existence of currently active brain metastasis.
3. HIV infection, active Hepatitis B or C infection, or active infections requiring oral or intravenous antibiotics or that can cause a severe disease and pose a severe danger to lab personnel working on patients' blood or tissue. If positive test results are not indicative of an active infection, patients can be included.
4. Treatment with excluded therapy per protocol
5. Previous extensive radiotherapy to the lung or liver during the last 4 months prior to lymphodepletion regimen.
6. The patient has cardiac conditions defined per protocol
7. Patients with prior stem cell transplantation or solid organ transplantation.
8. The patient has concurrent severe and/or uncontrolled medical disease that could compromise participation in the study
9. Active diverticulitis, intra-abdominal abscess, gastrointestinal obstruction, abdominal carcinomatosis or other known risk factors for bowel perforation.
10. History of other malignancies (except for adequately treated basal or squamous cell carcinoma or carcinoma in situ) within the last 3 years.
11. The patient is pregnant or is breastfeeding.
12. Serious autoimmune disease per protocol
13. History of hypersensitivity to cyclophosphamide, fludarabine or IL-2.
14. Immunosuppression, not related to prior treatment for malignancy.
15. History of or current immunodeficiency disease or prior treatment compromising immune function at the discretion of the treating physician.
16. Patients with Grade 3 or higher immune-related toxicities related to prior checkpoint inhibitors

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2021-09-22 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (Safety and tolerability) of IMA101 alone or in combination with atezolizumab | up to 18 months

SECONDARY OUTCOMES:
Peripheral T-cell persistence (assessment of frequency of T-cells over time) | up to 18 months
Tumor response per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 and immune-related RECIST (irRECIST) | up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Cedrik Britten, M.D., Study Director — Immatics US, Inc.
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tsimberidou AM, Guenther K, Andersson BS, Mendrzyk R, Alpert A, Wagner C, Nowak A, Aslan K, Satelli A, Richter F, Kuttruff-Coqui S, Schoor O, Fritsche J, Coughlin Z, Mohamed AS, Sieger K, Norris B, Ort R, Beck J, Vo HH, Hoffgaard F, Ruh M, Backert L, Wistuba II, Fuhrmann D, Ibrahim NK, Morris VK, Kee BK, Halperin DM, Nogueras-Gonzalez GM, Kebriaei P, Shpall EJ, Vining D, Hwu P, Singh H, Reinhardt C, Britten CM, Hilf N, Weinschenk T, Maurer D, Walter S. Feasibility and Safety of Personalized, Multi-Target, Adoptive Cell Therapy (IMA101): First-in-Human Clinical Trial in Patients with Advanced Metastatic Cancer. Cancer Immunol Res. 2023 Jul 5;11(7):925-945. doi: 10.1158/2326-6066.CIR-22-0444. PMID 37172100
- [Derived] Fritsche J, Rakitsch B, Hoffgaard F, Romer M, Schuster H, Kowalewski DJ, Priemer M, Stos-Zweifel V, Horzer H, Satelli A, Sonntag A, Goldfinger V, Song C, Mahr A, Ott M, Schoor O, Weinschenk T. Translating Immunopeptidomics to Immunotherapy-Decision-Making for Patient and Personalized Target Selection. Proteomics. 2018 Jun;18(12):e1700284. doi: 10.1002/pmic.201700284. Epub 2018 Apr 10. PMID 29505699